CLINICAL TRIAL: NCT01255501
Title: A First in Man Randomized Placebo Controlled Study of Single Ascending Intravenous Doses of NI-0701 in Healthy Volunteers
Brief Title: First in Human Study of NI-0701 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Other Study IDs: NI-0701-01
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteers

ARMS (2):
- NI-0701 (Experimental)
  Interventions: Drug: NI-0701
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NI-0701
  Arms: NI-0701
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, pharmacodynamic and pharmacokinetic profiles of a novel therapeutic drug when administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Non smokers
* Able to adhere to study visits and protocol requirements

Exclusion Criteria:

* Any clinical safety laboratory measurements value > Grade 1 on WHO Toxicity Scale
* Established or recurrent history of allergic reactions

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Safety and tolerability of escalating single IV doses of NI-0701 in healthy volunteers

SECONDARY OUTCOMES:
NI-0701 Pharmacokinetic parameters in healthy volunteers
NI-0701 plasma pharmacodynamic effects upon NI-0701 single intravenous infusion
Pharmacodynamic effects of NI-0701 on Histamine skin-induced wheal and flare
Immunogenicity of NI-0701

CONTACTS AND LOCATIONS:
Overall Officials: John Lambert, MD, Principal Investigator — PXL
Locations (1):
- London, United Kingdom